CLINICAL TRIAL: NCT00525889
Title: A Phase I Trial of Proleukin and Rapamune in Recent-onset Type 1 Diabetes Mellitus (ITN018AI)
Brief Title: Proleukin and Rapamune in Type 1 Diabetes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Immune Tolerance Network (ITN) (Network)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DAIT ITN018AI
Record Dates: First submitted 2007-09-04; First posted 2007-09-06 (Estimated); Last update posted 2017-02-08 (Estimated); Status verified 2017-02

CONDITIONS: Diabetes Mellitus, Type 1
Keywords: diabetes; juvenile diabetes; type 1 diabetes; diabetes mellitus; recent onset; new onset
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus | interventions — Interleukin-2; aldesleukin; Sirolimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Rapamycin/IL-2 combination therapy (Experimental): IL-2 (Proleukin) was administered at 4.5 3 106 IU s.c., three times per week for 4 weeks for a total of 12 doses. Rapamycin (Rapamune or Sirolimus) was administered without a loading dose at 2 mg/day, with adjustments to maintain trough blood levels of 5-10 ng/mL for 3 months.
  Interventions: Drug: IL-2; Drug: Rapamycin

INTERVENTIONS:
Drug: IL-2 — Administered by subcutaneous injection at a dose of 4.5x10^6 IU/day, three times weekly for 28 days starting on day 0.
  Other Names: Proleukin
Drug: Rapamycin — Administered orally, initial daily dose of 2mg. At day 7, dose adjusted to achieve and maintain whole blood trough levels of 5-10 ng/ml.
  Other Names: Rapamune; Sirolimus

SUMMARY:
This is a phase I trial in individuals who have been diagnosed with type 1 diabetes within the previous 3-48 months. The study is testing whether two immune system modifying drugs are safe when used in combination and if they have immune altering effects that indicate they can halt the progression of type 1 diabetes progression.

DETAILED DESCRIPTION:
At the time of diagnosis with type 1 diabetes, 15-40% of beta cells may remain active and healthy in the pancreas, capable of producing insulin the body needs to regulate blood glucose levels. Because even small amounts of natural insulin production can decrease the long term effects of diabetes, it is essential that these cells are preserved.

This trial will test whether a combination of the drugs Proleukin (IL-2) and Rapamune (sirolimus) may be safely administered to recently diagnosed type 1 diabetes patients and whether it causes changes to the immune system that can halt the autoimmune destruction of the remaining beta cells. This drug combination has been found to be effective for long-term diabetes prevention in mouse models of type 1 diabetes.

This study is a phase I study for individuals 18-45 years of age who have been diagnosed with type 1 diabetes in the past 3-48 months. All participants will be treated with Proleukin (administered subcutaneously 3x per week) for 28 days and Rapamune (taken orally, daily) for 12 weeks. The study will last for 12 months, with additional follow-up of 24 months. The majority of study visits occur within the first 6 months. Mixed meal tolerance tests, in which participants take a milkshake-like drink and have blood sampled over a 2 or 4-hour period, will take place during an initial screening visit and three additional times during the first year. All participants will also receive intensive diabetes management designed to maintain stable blood glucose levels.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with type 1 diabetes (per ADA criteria) more than 3 but less than 48 months prior to enrollment;
* 18 to 45 years of age;and
* Positive for at least one islet cell autoantibody (GAD65-antibody, CA512-antibody and/or ICA).

Exclusion Criteria:

* Chronic use of glucocorticoids or other immunosuppressive ages 4 weeks before enrollment;
* History of recurrent infections, other autoimmune diseases, cardiac disease, cataracts or other chronic medical conditions that investigators believe could compromise participant safety;
* Females who are pregnant, lactating intend to get pregnant, or are unwilling to undergo pregnancy testing during the study;
* Males who intend to father a pregnancy during the first 6 months of the study; or
* Participation in another clinical study within the last 30 days.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 9 (Actual)
Dates: Start 2007-08; Primary Completion 2011-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Incidence and severity of adverse events and laboratory anomalies | through day 364

SECONDARY OUTCOMES:
AUC for C-peptide responses following MMTT | various
Frequency of severe hypoglycemia | various
Insulin dose in units per kilogram | various
HbA1c levels | various

CONTACTS AND LOCATIONS:
Overall Officials: Carla Greenbaum, MD, Principal Investigator — Benaroya Research Institute
Locations (3):
- United States (3):
  - Naomi Berrie Diabetes Center, Columbia University, New York, New York
  - Oregon Health Sciences University, Portland, Oregon
  - Benaroya Research Institute, Seattle, Washington

IPD SHARING:
Plan to Share IPD: Yes
Participant level data and additional relevant materials are available to the public in the Immunology Database and Analysis Portal (ImmPort). ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts.

REFERENCES:
- [Result] Long SA, Rieck M, Sanda S, Bollyky JB, Samuels PL, Goland R, Ahmann A, Rabinovitch A, Aggarwal S, Phippard D, Turka LA, Ehlers MR, Bianchine PJ, Boyle KD, Adah SA, Bluestone JA, Buckner JH, Greenbaum CJ; Diabetes TrialNet and the Immune Tolerance Network. Rapamycin/IL-2 combination therapy in patients with type 1 diabetes augments Tregs yet transiently impairs beta-cell function. Diabetes. 2012 Sep;61(9):2340-8. doi: 10.2337/db12-0049. Epub 2012 Jun 20. PMID 22721971
- [Derived] Prevel N, Allenbach Y, Klatzmann D, Salomon B, Benveniste O. Beneficial role of rapamycin in experimental autoimmune myositis. PLoS One. 2013 Nov 12;8(11):e74450. doi: 10.1371/journal.pone.0074450. eCollection 2013. PMID 24265670
- See also: National Institute of Allergy and Infectious Diseases (NIAID) website — https://www.niaid.nih.gov/
- See also: Division of Allergy, Immunology, and Transplantation (DAIT) website — https://www.niaid.nih.gov/about/dait
- See also: Immune Tolerance Network (ITN) website — http://www.immunetolerance.org
- Available data/document: Individual Participant Data Set: SDY565 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY565 — ImmPort study identifier is SDY565. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts available to the Public.
- Available data/document: Study protocol summary and -schematic, -design, -demographics, -lab tests, -mechanistic assays, and -files: SDY565 — http://www.immport.org/immport-open/public/study/study/displayStudyDetail/SDY565 — ImmPort study identifier is SDY565. ImmPort is a long-term archive of clinical and mechanistic data from DAIT-funded grants and contracts available to the Public.